CLINICAL TRIAL: NCT04664439
Title: Application of CT-derived Fractional Flow Reserve in Patients With Coronary Heart Disease After Drug-coated Balloon Intervention
Brief Title: Follow-up With CT-FFR in CHD Patients After DCB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Xue Yu, Vice Director of Cardiology Department, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-FFR after DCB
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Coronary; Ischemic
Keywords: CT-derived fractional flow reserve; drug-coated balloon
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-FFR (Experimental): The CCTA images of the patients in this group will be analyzed and the FFR values of the lesions will be measured using the indicated software. ICA will be determined according to the value of CTFFR.
  Interventions: Diagnostic Test: CT-FFR
- direct ICA (No Intervention): The patients will be submitted to undergoing ICA procedure according to the decision of the investigators.

INTERVENTIONS:
Diagnostic Test: CT-FFR — CCTA examination will be performed by qualified medical imaging technicians, and patients will be scanned with 256rows of CT, according to standard operating norms. The coronary artery physiological function evaluation software(Keya Medical Technology, Beijing, China)will be configured in the core laboratory in advance, and the relevant imaging analysts will be trained. The core laboratory will receive the CCTA inspection data and evaluate the CCTA image quality. According to the standard operation flow of the software specification, the CT-FFR analysis will be carried out on the images that meet the requirements, and the CT-FFR value of the lesions will be measured.
  Arms: CT-FFR

SUMMARY:
In recent years, based on CCTA data, CT-derived fractional flow reserve (CT-FFR) developed by artificial intelligence and other technologies can provide both anatomical and functional information of coronary artery disease. Compared with CCTA alone, CT-FFR has a better ability to diagnose coronary ischemic lesions and can effectively reduce the need for unnecessary ICA, to predict revascularization more accurately.

DETAILED DESCRIPTION:
Drug-coated balloon (DCB) intervention is a non-drug treatment of coronary heart disease with the advantage of "no implantation". In recent years, it is more and more used in primary coronary artery disease. Timely detection of restenosis after DCB is very important to ensure the safety of patients. Invasive coronary angiography (ICA) is the "gold standard" to reflect coronary artery stenosis, but it is difficult to become a routine follow-up tool for surgical trauma, radiation exposure and other reasons, let alone for elderly patients.

Coronary artery computed tomography angiography (CCTA) can provide a variety of anatomical information such as the degree of coronary artery stenosis and the nature of plaques. It is a commonly used tool for non-invasive imaging diagnosis of coronary heart disease. However, because of its low diagnostic specificity and can not reflect the lesion-related myocardial ischemia, the positive rate of coronary heart disease and the rate of revascularization in patients undergoing ICA are low. In recent years, based on CCTA data, CT-derived fractional flow reserve (CT-FFR) developed by artificial intelligence and other technologies can provide both anatomical and functional information of coronary artery disease. A number of studies have shown that, compared with CCTA alone, CT-FFR has a better ability to diagnose coronary ischemic lesions and can effectively reduce the need for unnecessary ICA, to predict revascularization more accurately. Due to the absence of metal foreign body implantation, DCB intervention makes it possible for CT-FFR to be used in imaging evaluation after DCB. At present, there is no study on the use of CT-FFR in patients after DCB.

In this study, the self-developed CT-FFR based on artificial intelligence was used for the first time to analyze coronary artery lesions in patients after DCB, and to compare the guiding value of CT-FFR and simple CCTA in ICA and revascularization, in order to provide an ideal non-invasive imaging follow-up tool for elderly patients after DCB.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand the purpose of the test and sign the informed consent form.
2. 6-12 months after DCB for coronary heart disease, there is no contraindication of coronary artery CTA examination.
3. Non-target lesions of unplanned revascularization within 6 months.
4. According to the clinical manifestations and auxiliary examinations (such as EET, SPECT, CCTA), the attending doctor will make a comprehensive judgment on the patients who plan to undergo ICA.

Exclusion Criteria:

Patient exclusion criteria:

1. Previous coronary artery bypass (CABG) surgery, coronary artery stent implantation, artificial heart valve implantation, cardiac pacemaker or implantable defibrillator implantation.
2. Persistent or active symptoms of clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure (systolic blood pressure less than 90 mmHg), severe congestive heart failure (NYHA heart function III or IV) or acute pulmonary edema.
3. Acute myocardial infarction occurred within 7 days before selection.
4. Patients with other severe diseases are not suitable to participate in clinical trials, such as history of complex congenital heart disease, sick sinus syndrome, long QT syndrome, severe arrhythmia or tachycardia, severe asthma, severe or extremely severe chronic obstructive pulmonary disease, chronic renal dysfunction (serum creatinine level > 2.0mg / dl or creatinine clearance < 30ml/ Kg ·1.73m2).
5. Allergic to iodinated contrast medium.
6. Other serious allergic diseases such as allergic asthma.
7. Pregnancy or pregnancy status unknown.
8. Life expectancy is less than 6 months.
9. There are any factors that other researchers think are not suitable for selection or completion of this study.

   -

CCTA image exclusion criteria:

1. Obvious dislocation of coronary artery image.
2. CCTA images indicate that the reference vessel diameter of the stenotic segment is less than 2.0mm.
3. The image of coronary artery calcification accounting for more than 80% of the cross-sectional area of the lumen.
4. The standard deviation of CT value (SD value) of aortic root image was higher than that of 30HU.
5. Coronary artery occlusion.
6. The CT-FFR measurement can not be completed due to the quality problem of the image file.
7. The clinical trial could not be completed and no effective data were obtained due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of non-obstructive coronary heart disease in ICA examination | Clinical follow-up at 6 months after ICA or CT-FFR
  Proportion of non-obstructive coronary heart disease in ICA examination

SECONDARY OUTCOMES:
The rate of major adverse cardiac events (MACEs) | Clinical follow-up at 6 months after ICA or CT-FFR
  A composite endpoint of MACEs, including revascularization, non-fatal myocardial infarction, death and readmission for chest pain

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yu, MD, Study Chair — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, China